CLINICAL TRIAL: NCT04492514
Title: Mavrilimumab to Reduce Progression of Acute Respiratory Failure in COVID-19 Pneumonia and Systemic Hyper-inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kristin Hudock (Other)
Collaborators: Kiniksa Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Kristin Hudock, Assistant Professor of Medicine and Pediatrics, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IND 149353
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: COVID 19; SARS-CoV 2; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — mavrilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mavrilimumab (Experimental): Mavrilimumab Treatment infusion
  Interventions: Drug: Mavrilimumab
- Placebo (Placebo Comparator): Placebo infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mavrilimumab — Treatment infusion
  Other Names: KPL-301
  Arms: Mavrilimumab
Drug: Placebo — Placebo infusion
  Other Names: Control
  Arms: Placebo

SUMMARY:
The purpose of this prospective, Phase 2, multicenter, blinded, randomized placebo controlled study is to demonstrate that early treatment with mavrilimumab prevents progression of respiratory failure in patients with severe COVID-19 pneumonia and clinical and biological features of hyper-inflammation.

DETAILED DESCRIPTION:
This prospective, Phase 2, multi-center, blinded randomized placebo-controlled study is designed to demonstrate that early treatment with mavrilimumab prevents progression of respiratory failure in patients with severe COVID-19 pneumonia and clinical and biological features of hyper-inflammation.

The study population includes patients who have severe pneumonia, defined as hospitalization due to COVID-19 with abnormal chest imaging and SpO2 <92% on room air or requirement for supplemental oxygen.

Enrollment: The study will be performed in approximately 4 months total, starting from the first patient enrolled with enrollment expected to complete within 2 months.

Follow-up Period: The follow-up period is 60 days for each patient enrolled.

A total of 60 patients will be randomized using 1:1 allocation ratio: 30 subjects will receive mavrilimumab, and 30 subjects will receive placebo infusion. The investigator, clinical team, and subject will be blinded to treatment assignment.

Participants will be identified by regular review of hospitalized COVID 19 patients to evaluate for inclusion and exclusion criteria. Participants will then be approached in this standard manner by study investigator and/or coordinator/research nurse.

Research interventions will take place in the hospital in accordance with privacy standards.

The study team in informed on all study procedures and requirements with daily meetings and the opportunity to continuously update through secure channels.

In this multicenter consortium of 4 academic centers, each participating site will have their own IND for patients enrolled at their site. Data collection will occur at each of the 4 academic centers. Data analysis and randomization scheme will be performed by the Cleveland Clinic C5 Research, data analysis, and randomization scheme will be performed by one site, Cleveland Clinic C5 Research.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (must meet all):

1. Written informed consent must be obtained before any assessment is performed
2. Documented COVID19 pneumonia defined as positive SARS-CoV2 test AND abnormalities/ infiltrates on chest x-ray or computed tomography AND active fever or documented fever within 24-48 hours or ongoing anti-pyretic use to suppress fever
3. Hypoxia (Room air SpO2 <92% or requirement for supplemental oxygen)
4. Increased serum inflammatory marker (CRP > 5 mg/dL)
5. Severity of disease warrants inpatient hospitalization

Exclusion Criteria:

1. Onset of COVID-19 symptoms >14 days
2. Age < 18 years-old
3. Hospitalized >7 days
4. Mechanically ventilated
5. Serious concomitant illness which in the opinion of the investigator precludes the patient from enrolling in the trial, including (but not limited to):

   * History of immunodeficiency (congenital or acquired)
   * Neutropenia (absolute neutrophil count <1,500/mm3)
   * History of solid-organ or bone marrow transplant
   * History of current systemic autoimmune or autoinflammatory disease(s) requiring systemic immune-modulating drugs
   * History of myeloproliferative disorder or active malignancy receiving cytotoxic chemotherapy
   * Pre-existing severe pulmonary disease (i.e. steroid dependent asthma, COPD on home oxygen, or other restrictive/obstructive lung disease requiring home oxygen)
   * Pre-existing severe left ventricular systolic dysfunction (i.e. LVEF <35%)
   * Known or suspected active tuberculosis (TB), latent TB, or history of incompletely treated TB or at high risk for latent TB (from exposure or prior incarceration)
   * History of active or latent viral hepatitis (i.e. Hepatitis B or C)
   * Concomitant uncontrolled systemic bacterial or fungal infection
   * Concomitant viral infection other than COVID-19 (e.g. Influenza, other respiratory viruses)
   * History of chronic liver disease with portal hypertension
   * History of end-stage renal disease on chronic renal replacement therapy
6. Recent treatment with cell-depleting biological therapies (e.g., anti- CD20) within 12 months, cell-depleting biological therapies (such as anti-tumor necrosis factor [TNF], anakinra, anti-Interleukin [IL]-6 receptor [e.g. tocilizumab], or abatacept) within 8 weeks (or 5 half-lives, whichever is longer), treatment with alkylating agents within 12 weeks, treatment with cyclosporine A, azathioprine, cyclophosphamide, or mycophenolate mofetil (MMF) within 4 weeks
7. Recent treatment with intramuscular live (attenuated) vaccine within 4 weeks
8. Chronic or recent corticosteroid use > 10 mg/day
9. Pregnant. Breast-feeding women are eligible with the decision to continue or discontinue breast-feeding during therapy taking into account the risk of infant exposure, the benefits of breast-feeding to the infant, and benefits of treatment to the mother
10. Enrolled in another investigational study using immunosuppressive therapy
11. Known hypersensitivity to mavrilimumab or any of its excipients
12. In the opinion of the investigator, unable to comply with the requirements to participate in the study
13. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of investigational drug. Such methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
    * Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Hudock, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cremer PC, Abbate A, Hudock K, McWilliams C, Mehta J, Chang SY, Sheng CC, Van Tassell B, Bonaventura A, Vecchie A, Carey B, Wang Q, Wolski KE, Rajendram P, Duggal A, Wang TS, Paolini JF, Trapnell BC; MASH-COVID study group. Mavrilimumab in patients with severe COVID-19 pneumonia and systemic hyperinflammation (MASH-COVID): an investigator initiated, multicentre, double-blind, randomised, placebo-controlled trial. Lancet Rheumatol. 2021 Jun;3(6):e410-e418. doi: 10.1016/S2665-9913(21)00070-9. Epub 2021 Mar 17. PMID 33754144

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mavrilimumab | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 participant was enrolled at our site and this individual received Mavrilimumab. We did not enroll any patients into the placebo group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mavrilimumab | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (0) |  | 66 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Alive and Off Oxygen at 14 Days
Description: Number of subjects alive and off of oxygen
Time Frame: 14 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Mavrilimumab | Placebo
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

2. Secondary Outcome: Proportion of Subjects Alive and Without Respiratory Failure at 28 Days
Description: Number of subjects alive and without respiratory failure
Time Frame: 28 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Mavrilimumab | Placebo
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 60 days
Description: Daily assessment and chart review with routine labs while inpatient. Virtual telehealth assessment on day 14, 21, 28, and 60.
Arm/Group | Mavrilimumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mavrilimumab (N=1) | Placebo (N=0)
Chest Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — dry cough, chest congestion, runny nose, sore throat, headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT04492514/Prot_SAP_000.pdf